CLINICAL TRIAL: NCT06831396
Title: Communication in Children with or Without Biomedical Conditions: Speech and Language Profile, Related Outcomes and Articulation Treatment with Ultrasound
Brief Title: Effectiveness of Ultrasound-Aided Articulation Therapy for Children with Speech Sound Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Yiu Oi Yan, Principal Investigator, The University of Hong Kong
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UW 23-522; HKU/HA HKW IRB (Other: Hong Kong Hospital Authority); Central IRB (Other: Hong Kong Hospital Authority)
Record Dates: First submitted 2025-02-14; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: ENT System; Cleft Palate Children; Brain Tumor
Keywords: Speech and Language; Children; Treatment; Ultrasound
MeSH Terms: conditions — Brain Neoplasms; Speech; Language

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the treatment group (n=30) or the waitlist control group (n=30), and stratified to the groups by disorders, age and gender whenever possible. The treatment group will receive the intervention immediately, while the waitlist control group will not receive the treatment until the initial treatment group has completed the study. This design allows for a comparison of outcomes between the treatment and control groups, while also ensuring that all participants have the opportunity to receive the treatment.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- case group (Other): Dose comparison (same intervention)
  Interventions: Behavioral: Dose comparison (same intervention)
- Control Group (Other): Dose comparison (same intervention)
  Interventions: Behavioral: Dose comparison (same intervention)

INTERVENTIONS:
Behavioral: Dose comparison (same intervention) — The intervention under investigation is a motor-phonetic approach to articulation therapy, enhanced with ultrasound visual biofeedback (UVBF). The treatment group will receive the intervention immediately, while the waitlist control group will receive treatment after the initial group completes the study. This design allows for comparative outcome assessments between both groups, ensuring that all participants ultimately receive treatment.

SUMMARY:
The study is a prospective randomized controlled procedure to investigate the effect of ultrasound in articulation training and also the effect of treatment intensity in this mode of therapy. Targeted subjects are children with brain tumor or cleft palate with articulation errors which visualization of lingual movement using ultrasound may facilitate their acquisition of the sounds misarticulated. Subjects would be randomized to two groups of high and low treatment intensity, with stratification to the groups by disorders, age and gender whenever possible. Participants will be randomly assigned to either the treatment group or a waitlist control group in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* No syndromes or obvious dysmorphic features; No language disorders associated with biomedical conditions (e.g., cerebral palsy, autism spectrum disorder); No oronasal fistula identified in oral examination or diagnosed velopharyngeal insufficiency; Hearing thresholds between 0 to 25 dB in at least one ear, with no hearing loss exceeding 50 dB in the other; Cantonese as the first language

Exclusion Criteria:

* Subjects with syndrome, speech or language disorder associated with biomedical conditions (e.g. cerebral palsy, autism spectrum disorder), hearing threshold higher than 25dB in one ear and hearing loss with more than 50dB in another ear would be excluded from the study. Participants would be excluded fromthe study if they have other planned surgical intervention during the study period.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Standardized perceptual speech assessment (HKCAT/C-CSAT) | Week0, Week 4, Week 8, Week 16
20-item probe list | Week0, Week4, Week8, Week16
treated and untreated word lists | Week1-3, Week4

SECONDARY OUTCOMES:
Intelligibility in Context Scale (ICS): Traditional Chinese | Week1, Week4, Week 8, Week 16
PedsQL TM (Pediatric Quality of Life Inventory TM) | Week 0, Week 4, Week 8,Week 16
Strengths and Difficulties Questionnaire (SDQ) | Week 0, Week4, Week 8, Week16
Parental Stress Scale (PSS) | Week0, Week 4, Week 8, Week 16
The Hong Kong Cantonese Articulation Test (HKCAT) | Week0
Cantonese-Cleft Speech Assessment Tool (C-CSAT) | Week0
The Hong Kong Cantonese Oral Language Scale (HKCOLAS) | Week0
CLEFT-Q Speech Function Scale, Cantonese version | Week0

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Children's Hospital and Child Assessment Centre of The Duchess of Kent Children's Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Hitchcock ER, Swartz MT, Lopez M. Speech Sound Disorder and Visual Biofeedback Intervention: A Preliminary Investigation of Treatment Intensity. Semin Speech Lang. 2019 Mar;40(2):124-137. doi: 10.1055/s-0039-1677763. Epub 2019 Feb 22. PMID 30795023
- [Background] Morgan AT, Murray E, Liegeois FJ. Interventions for childhood apraxia of speech. Cochrane Database Syst Rev. 2018 May 30;5(5):CD006278. doi: 10.1002/14651858.CD006278.pub3. PMID 29845607
- [Background] Alighieri C, Van Lierde K, De Caesemaeker AS, Demuynck K, Bruneel L, D'haeseleer E, Bettens K. Is High-Intensity Speech Intervention Better? A Comparison of High-Intensity Intervention Versus Low-Intensity Intervention in Children With a Cleft Palate. J Speech Lang Hear Res. 2021 Sep 14;64(9):3398-3415. doi: 10.1044/2021_JSLHR-21-00189. Epub 2021 Aug 25. PMID 34433000
- [Background] Alighieri C, Van Lierde K, Cammu H, Vanoost L, Bettens K. The retrospective acceptability of high intensity versus low intensity speech intervention in children with a cleft palate: A qualitative study from the parents' point of view using the Theoretical Framework of Acceptability. Int J Lang Commun Disord. 2023 Mar;58(2):326-341. doi: 10.1111/1460-6984.12788. Epub 2022 Oct 3. PMID 36189983
- [Background] Allen MM. Intervention efficacy and intensity for children with speech sound disorder. J Speech Lang Hear Res. 2013 Jun;56(3):865-77. doi: 10.1044/1092-4388(2012/11-0076). Epub 2012 Dec 28. PMID 23275415
- [Background] Cleland J, Crampin L, Campbell L, Dokovova M. Protocol for SonoSpeech Cleft Pilot: a mixed-methods pilot randomized control trial of ultrasound visual biofeedback versus standard intervention for children with cleft lip and palate. Pilot Feasibility Stud. 2022 Apr 27;8(1):93. doi: 10.1186/s40814-022-01051-x. PMID 35477444
- [Background] Sugden E, Lloyd S, Lam J, Cleland J. Systematic review of ultrasound visual biofeedback in intervention for speech sound disorders. Int J Lang Commun Disord. 2019 Sep;54(5):705-728. doi: 10.1111/1460-6984.12478. Epub 2019 Jun 10. PMID 31179581
- [Background] Gibson T, Lee SAS. Use of ultrasound visual feedback in speech intervention for children with cochlear implants. Clin Linguist Phon. 2021 May 4;35(5):438-457. doi: 10.1080/02699206.2020.1792996. Epub 2020 Jul 17. PMID 32677475
- [Background] Marchant J, McAuliffe MJ, Huckabee ML. Treatment of articulatory impairment in a child with spastic dysarthria associated with cerebral palsy. Dev Neurorehabil. 2008 Jan-Mar;11(1):81-90. doi: 10.1080/17518420701622697. PMID 17943504
- [Background] Nordberg A, Miniscalco C, Lohmander A, Himmelmann K. Speech problems affect more than one in two children with cerebral palsy: Swedish population-based study. Acta Paediatr. 2013 Feb;102(2):161-6. doi: 10.1111/apa.12076. Epub 2012 Nov 27. PMID 23186066
- [Background] Hayden DA, Square PA. Motor Speech Treatment Hierarchy: a systems approach. Clin Commun Disord. 1994 Sep;4(3):162-74. PMID 7994291
- [Background] Pennington L, Roelant E, Thompson V, Robson S, Steen N, Miller N. Intensive dysarthria therapy for younger children with cerebral palsy. Dev Med Child Neurol. 2013 May;55(5):464-71. doi: 10.1111/dmcn.12098. Epub 2013 Feb 26. PMID 23441834
- [Background] Pennington L, Miller N, Robson S, Steen N. Intensive speech and language therapy for older children with cerebral palsy: a systems approach. Dev Med Child Neurol. 2010 Apr;52(4):337-44. doi: 10.1111/j.1469-8749.2009.03366.x. Epub 2009 Sep 16. PMID 19758364
- [Background] Fox CM, Boliek CA. Intensive voice treatment (LSVT LOUD) for children with spastic cerebral palsy and dysarthria. J Speech Lang Hear Res. 2012 Jun;55(3):930-45. doi: 10.1044/1092-4388(2011/10-0235). Epub 2012 Jan 9. PMID 22232407
- [Background] Morgan AT, Vogel AP. A Cochrane review of treatment for dysarthria following acquired brain injury in children and adolescents. Eur J Phys Rehabil Med. 2009 Jun;45(2):197-204. Epub 2009 Jan 21. PMID 19156018
- [Background] Pennington L, Parker NK, Kelly H, Miller N. Speech therapy for children with dysarthria acquired before three years of age. Cochrane Database Syst Rev. 2016 Jul 18;7(7):CD006937. doi: 10.1002/14651858.CD006937.pub3. PMID 27428115
- [Background] Michi K, Yamashita Y, Imai S, Suzuki N, Yoshida H. Role of visual feedback treatment for defective /s/ sounds in patients with cleft palate. J Speech Hear Res. 1993 Apr;36(2):277-85. doi: 10.1044/jshr.3602.277. PMID 8487520
- [Background] Lee AS, Law J, Gibbon FE. Electropalatography for articulation disorders associated with cleft palate. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):CD006854. doi: 10.1002/14651858.CD006854.pub2. PMID 19588407
- [Background] Alighieri C, Bettens K, Bruneel L, Perry J, Hens G, Van Lierde K. One Size Doesn't Fit All: A Pilot Study Toward Performance-Specific Speech Intervention in Children With a Cleft (Lip and) Palate. J Speech Lang Hear Res. 2022 Feb 9;65(2):469-486. doi: 10.1044/2021_JSLHR-21-00405. Epub 2022 Jan 12. PMID 35021015
- [Background] Bessell A, Sell D, Whiting P, Roulstone S, Albery L, Persson M, Verhoeven A, Burke M, Ness AR. Speech and language therapy interventions for children with cleft palate: a systematic review. Cleft Palate Craniofac J. 2013 Jan;50(1):e1-e17. doi: 10.1597/11-202. Epub 2012 Mar 20. PMID 22433039
- [Background] Lane H, Harding S, Wren Y. A systematic review of early speech interventions for children with cleft palate. Int J Lang Commun Disord. 2022 Jan;57(1):226-245. doi: 10.1111/1460-6984.12683. Epub 2021 Nov 12. PMID 34767284
- [Background] Yeung NC, Lau JT, Yu XN, Chu Y, Shing MM, Leung TF, Li CK, Fok TF, Mak WW. Psychometric properties of the Chinese version of the Pediatric Quality Of Life Inventory 4.0 Generic Core scales among pediatric cancer patients. Cancer Nurs. 2013 Nov-Dec;36(6):463-73. doi: 10.1097/NCC.0b013e31827028c8. PMID 23059765
- [Background] Lau JT, Yu XN, Chu Y, Shing MM, Wong EM, Leung TF, Li CK, Fok TF, Mak WW. Validation of the Chinese version of the Pediatric Quality of Life Inventory (PedsQL) Cancer Module. J Pediatr Psychol. 2010 Jan-Feb;35(1):99-109. doi: 10.1093/jpepsy/jsp035. Epub 2009 May 6. PMID 19420227
- [Background] Nicola K, Watter P. Health-related quality of life from the perspective of children with severe specific language impairment. Health Qual Life Outcomes. 2015 Aug 14;13:127. doi: 10.1186/s12955-015-0326-1. PMID 26268357
- [Background] Varni JW, Limbers CA, Burwinkle TM. Impaired health-related quality of life in children and adolescents with chronic conditions: a comparative analysis of 10 disease clusters and 33 disease categories/severities utilizing the PedsQL 4.0 Generic Core Scales. Health Qual Life Outcomes. 2007 Jul 16;5:43. doi: 10.1186/1477-7525-5-43. PMID 17634123
- [Background] Schmitt LC, Paterno MV, Huang S. Validity and internal consistency of the international knee documentation committee subjective knee evaluation form in children and adolescents. Am J Sports Med. 2010 Dec;38(12):2443-7. doi: 10.1177/0363546510374873. Epub 2010 Aug 30. PMID 20805408
- [Background] Varni JW, Seid M, Rode CA. The PedsQL: measurement model for the pediatric quality of life inventory. Med Care. 1999 Feb;37(2):126-39. doi: 10.1097/00005650-199902000-00003. PMID 10024117
- [Background] Gomersall T, Spencer S, Basarir H, Tsuchiya A, Clegg J, Sutton A, Dickinson K. Measuring quality of life in children with speech and language difficulties: a systematic review of existing approaches. Int J Lang Commun Disord. 2015 Jul;50(4):416-35. doi: 10.1111/1460-6984.12147. Epub 2015 Jan 29. PMID 25630911
- [Background] Markham C, Dean T. Parents' and professionals' perceptions of Quality of Life in children with speech and language difficulty. Int J Lang Commun Disord. 2006 Mar-Apr;41(2):189-212. doi: 10.1080/13682820500221485. PMID 16546895
- [Background] Feeney R, Desha L, Khan A, Ziviani J. Contribution of speech and language difficulties to health-related quality-of-life in Australian children: A longitudinal analysis. Int J Speech Lang Pathol. 2017 Apr;19(2):139-152. doi: 10.3109/17549507.2016.1151935. Epub 2016 Apr 4. PMID 27063693
- [Background] Lancaster HS, Lien KM, Chow JC, Frey JR, Scherer NJ, Kaiser AP. Early Speech and Language Development in Children With Nonsyndromic Cleft Lip and/or Palate: A Meta-Analysis. J Speech Lang Hear Res. 2019 Dec 13;63(1):14-31. doi: 10.1044/2019_JSLHR-19-00162. Print 2020 Jan 22. PMID 31841365
- [Background] Boyce JO, Kilpatrick N, Reilly S, Da Costa A, Morgan AT. Receptive and expressive language characteristics of school-aged children with non-syndromic cleft lip and/or palate. Int J Lang Commun Disord. 2018 Sep;53(5):959-968. doi: 10.1111/1460-6984.12406. Epub 2018 Jul 3. PMID 29968398
- [Background] Feragen KB, Saervold TK, Aukner R, Stock NM. Speech, Language, and Reading in 10-Year-Olds With Cleft: Associations With Teasing, Satisfaction With Speech, and Psychological Adjustment. Cleft Palate Craniofac J. 2017 Mar;54(2):153-165. doi: 10.1597/14-242. Epub 2015 Jun 29. PMID 26120883
- [Background] Klinto K, Salameh EK, Lohmander A. Verbal competence in narrative retelling in 5-year-olds with unilateral cleft lip and palate. Int J Lang Commun Disord. 2015 Jan-Feb;50(1):119-28. doi: 10.1111/1460-6984.12127. Epub 2014 Sep 11. PMID 25208601
- [Background] Chapman KL. The relationship between early reading skills and speech and language performance in young children with cleft lip and palate. Cleft Palate Craniofac J. 2011 May;48(3):301-11. doi: 10.1597/08-213. Epub 2010 Aug 17. PMID 20815721
- [Background] Collett BR, Leroux B, Speltz ML. Language and early reading among children with orofacial clefts. Cleft Palate Craniofac J. 2010 May;47(3):284-92. doi: 10.1597/08-172.1. PMID 20426677
- [Background] Flynn T, Moller C, Jonsson R, Lohmander A. The high prevalence of otitis media with effusion in children with cleft lip and palate as compared to children without clefts. Int J Pediatr Otorhinolaryngol. 2009 Oct;73(10):1441-6. doi: 10.1016/j.ijporl.2009.07.015. Epub 2009 Aug 25. PMID 19709760
- [Background] Sell D, Harding A, Grunwell P. GOS.SP.ASS.'98: an assessment for speech disorders associated with cleft palate and/or velopharyngeal dysfunction (revised). Int J Lang Commun Disord. 1999 Jan-Mar;34(1):17-33. doi: 10.1080/136828299247595. PMID 10505144
- [Background] John A, Sell D, Sweeney T, Harding-Bell A, Williams A. The cleft audit protocol for speech-augmented: A validated and reliable measure for auditing cleft speech. Cleft Palate Craniofac J. 2006 May;43(3):272-88. doi: 10.1597/04-141.1. PMID 16681400
- [Background] Taylor OD, Ware RS, Weir KA. Speech pathology services to children with cancer and nonmalignant hematological disorders. J Pediatr Oncol Nurs. 2012 Mar-Apr;29(2):98-108. doi: 10.1177/1043454212438963. PMID 22472483
- [Background] Simms MD. Language disorders in children: classification and clinical syndromes. Pediatr Clin North Am. 2007 Jun;54(3):437-67, v. doi: 10.1016/j.pcl.2007.02.014. PMID 17543904
- [Background] Snowling MJ, Bishop DV, Stothard SE, Chipchase B, Kaplan C. Psychosocial outcomes at 15 years of children with a preschool history of speech-language impairment. J Child Psychol Psychiatry. 2006 Aug;47(8):759-65. doi: 10.1111/j.1469-7610.2006.01631.x. PMID 16898989
- See also: 9Patients Profile Treated by Speech-language therapy Service, with Emphasis on Language in a Children's Hospital — https://www.thieme-connect.de/products/ejournals/abstract/10.1055/s-0034-1388959